CLINICAL TRIAL: NCT04336917
Title: Ultrasound Guided Rhomboid Intercostal and Subserratus Plane Block in Breast Cancer Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Breast Cancer-RISS
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer Surgery; Postoperative Analgesia
Keywords: Rhomboid intercostal and subserratus plane block
MeSH Terms: interventions — Anesthetics, Local; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Prospective study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Rhomboid Intercostal and Subserratus Plane Block (Active Comparator): In addition to routine standard perioperative and postoperative analgesic protocol participants will recieve Rhomboid Intercostal and Subserratus Plane Block under ultrasound guidence at the end of the surgery.
  Interventions: Drug: Rhomboid Intercostal and Subserratus Plane Block with local anesthetic
- Control Group (No Intervention): Routine standard perioperative and postoperative analgesic protocol will be given.

INTERVENTIONS:
Drug: Rhomboid Intercostal and Subserratus Plane Block with local anesthetic — Local anesthetic will be injected in the tissue planes between the rhomboid and the intercostal muscles and the serratus anterior and external intercostal muscles with ultrasound guidence.
  Other Names: 40 mL of bupivacaine/lidocaine mixture
  Arms: Group Rhomboid Intercostal and Subserratus Plane Block

SUMMARY:
Postoperative analgesia after breast cancer surgery is a challenge for anesthesiologists due to the complex innervation of the breast. Interfascial plane blocks of the chest are gaining widespread popularity with the introduction of ultrasonography into the regional anesthesia practice. We aimed to investigate the efficacy of Rhomboid intercostal and subserratus plane block (RISS) for postoperative analgesia in patients undergoing breast cancer surgery.

DETAILED DESCRIPTION:
This prospective randomized controlled trial will be carried out on female patients who scheduled for breast cancer surgery. Our hypotesis is that this new interfascial plane block technique will able to provide postoperative analgesia in breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-85 years and ASA physiological score I-III who undergone breast cancer surgery

Exclusion Criteria:

* Patients refused to participate.
* Patients with known or suspected allergy to the used medication.
* Patients with psychiatric-neurological disorders that may affect pain perception,
* Patients regularly taking antipsychotics and antidepressants.
* Patients with potential risk of coagulopathy.
* Uncooperative patients.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative opiod consumption | The first 24 hours postoperatively
  Opioid consumptions for both group will be recorded.

SECONDARY OUTCOMES:
Postoperative pain scores | The first 24 hours postoperatively
  Postoperative pain will be assessed using a Numeric Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst imaginable pain).The NRS will be recorded in postoperative unit and in ward at first hour and at 2th, 6th, 12th and 24 th hour.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Kozanhan, M.D., Principal Investigator — SBÜ Konya EAH
Locations (1):
- Konya Education and Training Hospital, Konya, Turkey (Türkiye)